CLINICAL TRIAL: NCT01412073
Title: A Randomized Trial to Determine the Best Strategy for the Control of Blood Loss at Elective Caesarean Section
Brief Title: Control of Blood Loss During Caesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Waleed El-khayat, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 582011
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Complications; Cesarean Section
Keywords: caesarean section, intrapartum haemorrhage
MeSH Terms: interventions — Oxytocin; Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- oxytocin bolus (Active Comparator): 5 IU bolus iv over 3 minutes after delivery of the baby Operative blood loss will be estimated in theatre based on the volume in the suction bottle and the weight of swabs used. We will record blood loss up until the time the woman will be discharged from the theatre recovery ward.
  Hemoglobin level and haematocrit value will be done as follow:-
  1. After admission of each case in the pre-operative period.
  2. Immediately post- operative.
  3. 24 hours post- operative.
  Interventions: Drug: oxytocin
- oxytocin bolus & oxytocin infusion (Active Comparator): 5 IU oxytoxin bolus over 3 minutes and 30 IU oxytocin infusion in 500 ml 0.9% saline over 4 hours after delivery of the baby
  Interventions: Drug: oxytocin
- misoprostol intrauterine (Active Comparator): misoprostol 800 micrograms intrauterine, placed manually on the bottom of the uterine cavity after delivery of the placenta and cleaning of the cavity
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: oxytocin — group I : oxytocin 5 IU bolus over 3 minutes after delivery of the baby group II : oxytocin 5 IU bolus over 3 minutes after delivery of the baby and oxytocin infusion in 500 ml 0.9% saline over 4 hours
  Other Names: syntocinon
  Arms: oxytocin bolus; oxytocin bolus & oxytocin infusion
Drug: Misoprostol — misoprostol intrauterine 800 microgram placed intrauterine after delivery of the baby & the placenta
  Other Names: cytotec
  Arms: misoprostol intrauterine

SUMMARY:
trial of 3 protocols to determine the best one to control blood loss during caesarean section

DETAILED DESCRIPTION:
The study population will be divided into 3 groups each containing 200 women:

Group (A): 200 patients will receive 5-IU oxytocin bolus over 3 minutes after delivery of the baby.

Group (B): 200 patients will receive 5-IU oxytocin bolus over 3 minutes and 30-IU oxytocin infusion in 500 ml 0.9 % saline over 4 hours after delivery of the baby.

Group (C): 200 patients will receive misoprostol 800 micrograms intrauterine, placed manually on the bottom of the uterine cavity after delivery of the placenta and cleaning of the cavity.

Operative blood loss will be estimated in theatre based on the volume in the suction bottle and the weight of swabs used. We will record blood loss up until the time the woman will be discharged from the theatre recovery ward.

Hemoglobin level and haematocrit value will be done as follow:-

1. After admission of each case in the pre-operative period.
2. Immediately post- operative.
3. 24 hours post- operative.

ELIGIBILITY:
Inclusion Criteria:

* Patients booked for elective cesarean section.
* Singleton pregnancies.
* Primigravida or multipara ,first cesarean section or previous .

Exclusion Criteria:

* Patients with obstetric hemorrhage.
* Uterine laceration.
* Placenta previa.
* Blood dyscrasias.
* Large fibroids.
* Multiple pregnancy.
* Pre-eclampsia.
* Marked maternal anemia.
* Previous history of PPH.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
amount of blood loss | 12 month

SECONDARY OUTCOMES:
Haemoglobin % and haematocrit value | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Waleed M El-khayat, M.D., Study Director — Lecturer of Obstetrics & Gynecology , Faculty of medicine, Cairo University
Locations (1):
- faculty of medicine , Cairo University, Cairo, Cairo Governorate, Egypt